CLINICAL TRIAL: NCT01779245
Title: The Impact of a Calcium Supplementation on Lipid Metabolism During Exercise.
Brief Title: Effect of High-calcium Intake on Substrate Metabolism During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 32AN3
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Lipid Metabolism
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): A chocolate milkshake with a normal calcium content will be consumed daily (235 kcal; 13 g protein; 42 g carbohydrate; 1 g fat, 400 mg calcium per serving).
  Interventions: Dietary Supplement: Placebo
- High-Calcium (Experimental): A chocolate milkshake with a high calcium content will be consumed daily (235 kcal; 13 g protein; 42 g carbohydrate; 1 g fat, 1400 mg calcium per serving).
  Interventions: Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Calcium — Milk-extracted calcium supplement will be used to modulate the calcium content of the milkshakes used.
  Arms: High-Calcium
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
A high-calcium intake can accelerate fat loss under energy-restricted diets. Part of this may be due to a shift in substrate metabolism where there is an increase in the rate of fat oxidation. However, whether high-calcium intake can influence substrate metabolism during exercise is not known. Accordingly, we aim to investigate the effect of 2 weeks of high-calcium intake on substrate metabolism during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (moderate-vigorous exercise >3 time per week)
* Male
* 18-40 yrs of age

Exclusion Criteria:

* Smoker
* Known Food Allergies
* Metabolic disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Substrate metabolism | 60 s samples every 3 min for 15 min
  Substrate metabolism will be assessed by the respiratory exchange ratio (rate of carbon dioxide production/rate of oxygen consumption) from samples of expired gas collected during the first 15 minutes of an incremental cycling test.

SECONDARY OUTCOMES:
Plasma non-esterified fatty acid concentrations | Every 3 min for 15 min
  Non-esterified fatty acid concentrations will be determined from plasma samples collected during the first 15 minutes of an incremental cycling test to indicate fatty acid availability.
Plasma glycerol concentrations | Every 3 min for 15 min
  Glycerol concentrations will be determined from plasma samples collected during the first 15 minutes of an incremental cycling test as a marker of lipolysis.

OTHER OUTCOMES:
Serum parathyroid hormone concentration | Baseline (Pre-post 2 week supplementation)
  Parathyroid hormone concentrations will be determined at rest before and after supplementation periods as a indicator of calcium status.
Plasma glucose-dependent insulinotropic peptide concentration | Baseline (Pre-post 2 week supplementation)
  Glucose-dependent insulinotropic peptide concentrations will be determined at rest before and after supplementation periods as a potential mechanism of any changes in metabolism.
Plasma glucagon-like peptide-1 concentration | Baseline (Pre-post 2 week supplementation)
  Glucagon-like peptide-1 concentrations will be determined at rest before and after supplementation periods as a potential mechanism of any changes in metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom